CLINICAL TRIAL: NCT02359396
Title: Effects of Oral Administration of a Chinese Proprietary Medicine, MZRW on Tolerability, Exposure and Pharmacokinetics in Healthy Subjects
Brief Title: A Randomized, Open-label, Three-arm Study of MZRW on Tolerability, Exposure and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Chair Professor, Director of Clinical Division,, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKBU/FRG2/13-14/025
Record Dates: First submitted 2015-01-27; First posted 2015-02-10 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-02

CONDITIONS: Functional Constipation; Gastrointestinal Disorders
Keywords: Randomized open-label study; Chinese Herbal; Constipation/drug therapy
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5.0g of MZRW (Experimental): The participants will receive 5.0g of MZRW at 9 am .
  Interventions: Drug: MZRW
- 7.5g of MZRW (Experimental): The participants will receive 7.5g of MZRW at 9 am.
  Interventions: Drug: MZRW
- 10g of MZRW (Experimental): The participants will receive 10g of MZRW at 9 am.
  Interventions: Drug: MZRW

INTERVENTIONS:
Drug: MZRW — MZRWs is composed of Fructus Cannabis (HuoMaRen), Radix et Rhizoma Rhei (DaHuang), Radix Paeoniae Alba (BaiShao), Semen Armeniacae Amarum (KuXingRen), Fructus Aurantii Immaturus (ZhiShi) and Cortex Magnoliae Officinalis (HouPo). All MZRW granules will be prepared by PuraPharm International (H.K.) Limited. The entire manufacturing process, from authenticating the raw materials to the final products, is in strict compliance with the standards of Good Manufactory Practice (GMP) and Chinese Pharmacopoeia.

SUMMARY:
This is a randomized open-label, three-arm, phase 1 clinical study. The investigators aim to investigate a Chinese Proprietary Medicine, MZRW on its tolerability, system exposure and pharmacokinetics profile.

DETAILED DESCRIPTION:
This is a randomized, open-label, three-arm study. The participants will be enrolled and randomized in a ratio of 1:1:1 to receive 5.0g, 7.5g, 10g b.i.d. of MZRW at 9 am respectively. The study drug, MZRW will be administrated to the participants by site personnel after participants have fasted overnight for more than 8 hours and 6 hours after administration. Each participant will consume a standardized meal. In addition, the participants refrain from Semen Cannabis Sativae, Semen Pruni Armeniacae, Radix Paeoniae, Fructus Immaturus Citri Aurantii, Cortex Magnoliae and Radix et Rhizoma Rhei foods for 3 days before the study until completion of the study.

Blood samples (5 ml each) will be collected from the medial cubital vein into evacuated tubes containing heparin just before and at 0.25, 0.5, 1, 2, 4, 8, 12h after administration and were immediately centrifuged (1700g, 10 min). Plasma fractions were stored at -20°C until analysis. All study procedures conduct in accordance with the ethical principles of the Declaration of Helsinki, consistent with Good Clinical Practice guidelines, and approved by Hong Kong Baptist University Ethics Committee on the Use of Human Subjects for Teaching and Research. Subjects will be given their written informed consent before participating in the study. Urine samples (50 ml each) will be collected the day before the administration and at 0 to 3h, 3 to 6h, 6 to 9h and 9 to 12h after administration. Plasma and urine fractions will be stored at -80°C until analysis.

ELIGIBILITY:
Healthy voluteers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability among Three Doses of MZRW | 12 hours

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 12 hours
the changes of plasma concentrations of MZRW ingredients in different time points | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Xiang Bian, MD, Ph. D, Principal Investigator — School of Chinese Medicine, Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China